CLINICAL TRIAL: NCT02022592
Title: Comparison of Lormetazepam and Midazolam Used as Sedatives for Patients That Require Intensive Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Univ.-Prof. Dr. med. C. Spies, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LoveMi
Record Dates: First submitted 2013-12-12; First posted 2013-12-30 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Sedation in Intensive Care Unit Patients
Keywords: Sedation management; Midazolam; Lormetazepam; Intensive care unit
MeSH Terms: interventions — lormetazepam; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lormetazepam (Experimental): The patient is treated on ICU not longer than 2 days. Dosage requirements according to Summary of product characteristics (Sedalam®).
  Interventions: Drug: Lormetazepam
- Midazolam (Active Comparator): The patient is treated on ICU not longer than 2 days. Dosage requirements according to Summary of product characteristics (Midazolam-ratiopharm®, Midazolam-hameln®).
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Lormetazepam
  Arms: Lormetazepam
Drug: Midazolam
  Arms: Midazolam

SUMMARY:
A goal directed , demand-driven administration of sedative drugs is an integral part of every intensive care treatment. During long-term application of sedatives, Midazolam is the most commonly used sedative in Europe.

One major objective is the problem of oversedation and agitation during an intensive care treatment due to the lack of controllability of available substances.

The Love-Mi RCT investigates the clinical controllability of Midazolam versus the newly available intravenous drug Lormetazepam.

DETAILED DESCRIPTION:
Midazolam is almost exclusively metabolized intrahepatically. The methyl-group at position 1 of the imidazole ring is oxidized by liver enzymes. The product is a-OH-midazolam. This reaction is catalyzed by a p450-dependent oxidase in the liver.

Active a-OH-midazolam is inactivated by a biotransformation type II reaction after conjugation. The water soluble, conjugated midazolam can be excreted by the kidney.

During an intensive care treatment, the p450 dependent metabolization is known to be a "bottleneck of elimination" as many drugs are inactivated by this pathway.

As the phase II (glucuronidation) is non-saturable in practice - the phase I reaction limits the metabolic capacity. This leads to unpredictable prolongation of midazolam effects.

In contrast, Lormetazepam is glucuronized directly at its OH-group during a phase II reaction. Since the glucuronidation is non-saturable, Lormetazepam is metabolized with nearly constant kinetics even if repeatedly administered.

Due to the pharmacokinetics we hypothesize that Lormetazepam has an improved controllability compared to midazolam. As this leads to less frequent agitation and over-sedation, we hypothesize that there are multiple beneficial clinical outcomes for patients treated with lormetazepam instead of midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated ICU patients with the need for sedatives to achieve or maintain the intended target-RASS (surgical/ nonsurgical).
* Age ≥ 18 years
* Patients who are incapable of giving consent at study inclusion: Written informed consent by patient's legal representative or an independent medical consultant, patients give informed consent subsequent if they are capable.
* Patients who are able to give informed consent at study inclusion: Written informed consent by patients for planned postoperative prolonged ventilatory support who undergo heart surgery
* Consensable patients for inclusion: with necessary intubation with analgosedation

Exclusion Criteria:

* Any bolus administration of benzodiazepines until 72hrs before inclusion (except from premedication due to anaesthesia).
* Continuous administration of benzodiazepines within the last 7 days before start of study drug application
* Titration phase: No way that a target RASS between -3 and 0 can be determined by the attending physician
* Known drug intolerance or allergy against lormetazepam, midazolam or one of the additional components.
* Addictive disorder
* Increased intracranial pressure
* Acute intoxication with alcohol, analgesics, sedatives, antipsychotics (neuroleptics, anti-depressives, lithium).
* Patients with cerebrale Pathology, which changes the controllability of sedation or die consciousness (e.g. patients known mental retardation due to syndromatic disorders or an infantile brain damage)
* Patients with a suspected or secured hypoxic brain damage
* Patients with intracranial surgery during actual hospital care
* Tetraplegic patients
* Myasthenia Gravis
* Cerebellar or spinal Ataxia
* Moribund patients with an expected lifespan of less than 24 hours.
* Sickle cell anaemia
* Thallassemia
* Enzyme related disorders that are associated with a severe decreased activity of UDP-glucoronyltransferase (e.g. M. Crigler- Najjar)
* Chronic liver insufficiency CHILD C with MELD Score > 17 before access to intensive care unit
* Diagnosed propofol intolerance/anamnestic propofol infusion Syndrome
* Known depression/suicidality
* Pregnancy (positive beta-HCG test from urine or positive beta-HCG laboratory test from serum (in anuric patients the serum beta-HCG test is obliged) or lactation
* Woman of child-bearing potential who are not using a highly effective contraception (Pearl - Index <1) until 3 months after study inclusion and during this trial
* Referral following an order of official authorities (court order or administrative decision) according to German Drug Law (AMG)

  §40 (1) 4
* Participation in clinical trials according to the German Drug Law (AMG) 30 days to and during the study
* Local staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Controllability of sedation | Up to 50 hours
  Controllability of sedation is defined as the percentage share of measures where the actual depth of sedation (measured with the Richmond Agitation and Sedation Scale) (RASS)) matches the target depths of sedation. The individual sedation target is defined by the attending physician. . It will be measured until 5 days after terminationduring administration of study drug until 2 hours after its termination.

SECONDARY OUTCOMES:
SOFA (Sequential Organ Failure Assessment) | Up to 8 days
Pain-Scores | Up to 28 days
  NRS-V (Numeric Rating Scale -V) and FPS-R (Faces Pain Scale-Revised) and BPS (Behavioral Pain Scale) and BPS-NI (Non-Intubated BPS)
  according to German consensus guidelines
Anxiety-Score | Up to 28 days
  Faces Anxiety Scale score
Concurrent medication for Analgesia and Sedation | Up to 8 days
  dose/time.
Delirium-screening-Instruments | Up to 28 days
  CAM-ICU (Confusion Assessment Method for Intensive Care Unit) ICDSC ( Intensive Care Delirium Screening Checklist) Nu-DESC (Nursing Delirium Screening Scale)
Mortality | Up to 90 days
Duration of mechanical ventilation and weaning from mechanical ventilation | Up to 8 days
Length of intensive care unit stay | During intensive care unit stay, an average of 14 days
Length of hospital stay | During hospital stay, an average of 28 days
Follow-up treatment regarding Patient- Documentation-Management-System | During hospital stay, an average of 28 days
  Discharge Mode
Length of sedation | Up to 56 hours
  During administration of study drug until 8 hours after its termination.
Number of changes in target Richmond agitation sedation scale (RASS) | Up to 56 hours
  During administration of study drug
Wake-up-time | Up to 8 days
  During administration of study drug until 5 days after its termination
Deviation from target Richmond agitation sedation scale (RASS) | Up to 8 days
  During administration of study drug
Quality of Life | Up to 90 days
  Questionnaire designed to measure quality of life (EQ-5D-3L)
Cognition 1 | Up to 28 days
  Minimental State Examination (MMSE)
Cognition 2 | Up to 90 days
  Mehrfach-Wortschatz-Intelligenztest (MWT)
Posttraumatic stress disorder | Up to 90 days
  The Post-Traumatic Stress Syndrome 14-Questions Inventory
Bedside measurement of Acetylcholinesterase activity (U/gHb) | Up to 8 days
  The Acetylcholinesterase activity will be measured on every study day out of a blood sample (10µl); It will be measured until 5 days after termination of study drug.
Organ dysfunctions | Up to 8 days
  It will be measured until 5 days after termination of study drug.
Depth of sedation 1 | During the operation
  Depth of sedation is measured by Electroencephalography and Electromyography (only surgical patients in the Centers Charité and Gießen)
Depth of sedation 2 | Up to 3 days
  Depth of sedation 2 is measured by Electroencephalography and Electromyography (intensive care unit patients only Center Charité)
Photomotor reflex | Up to 8 days
  Photo motor reflex variations are measured by video pupillometry (only Center Charité)
Pain threshold measurement | Up to 3 days
  Automatic measurement of specific pain reflexes
micro ribonucleic acid (rna) | Up to 24 hours
  micro rna panel is analysed (only Center Charité)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Univ.- Prof., Study Chair — Charite University, Berlin, Germany; Gernot Marx, MD, Univ.-Prof., Study Director — University RWTH Aachen
Locations (3):
- Germany (3):
  - Clinic for Anesthesiology, Intensive Care Medicine and Painmanagement, Johann-Wolfgang-Goethe-University, Frankfurt, Frankfurt Am Main
  - Clinic for Operative Intensive Care Medicine and Intermediate Care, University of RWTH, Aachen
  - Department of Anesthesiology and Intensive Care Medicine, Charité - University Medicine, Berlin